CLINICAL TRIAL: NCT03912142
Title: Diagnosis of Obstetric Anal Sphincter Injuries (OASIs) Using Transperineal Ultrasound Scan (TPUS)
Status: Completed | Type: Observational
Sponsor: Lewisham and Greenwich NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 196995
Record Dates: First submitted 2017-03-08; First posted 2019-04-11 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Obstetric Anal Sphincter Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Three dimensional transperineal ultrasound: This is a single arm study. All women who delivered vaginally will be included in the study .
  The planned interventions are:
  Clinical vaginal and rectal examination Three dimensional transperineal ultrasound.
  Interventions: Diagnostic Test: three dimensional Transperineal Ultrasound Scan

INTERVENTIONS:
Diagnostic Test: three dimensional Transperineal Ultrasound Scan — Diagnostic test: three dimensional transperineal ultrasound scan
  Other Names: TPUS

SUMMARY:
It is common for women to sustain perineal trauma following their first vaginal delivery. Sometimes these can extend to the anal sphincter, and these are referred to as Obstetric Anal Sphincter Injuries (OASIs). Occasionally OASIs may not be detected at delivery. If these tears are missed they would not be repaired and this may lead to incontinence of wind (flatus) or of faeces, both of which can have a significant impact on quality of life. The investigators would like to establish whether a 3D ultrasound scan probe placed outside the vagina can identify the anal sphincter defects and to investigate whether the use of TPUS immediately after primary repair of OASIs is an useful tool to minimise an inadequate repair. The investigators would also like to look at changes that occur to the pelvic floor muscles during labour and to identify injuries to the pelvic floor muscle (levator ani) by ultrasound. Such injury to pelvic floor muscle is associated with vaginal prolapse.

DETAILED DESCRIPTION:
Following the first vaginal delivery 85% of women will sustain perineal trauma (1). Sometimes these can extend to the anal sphincter, and these are referred to as Obstetric Anal Sphincter Injuries (OASIs).

Occasionally OASIs may not be detected at delivery. If these tears are missed they would not be repaired and this may lead to incontinence of wind (flatus) or of faeces, both of which can have a significant impact on quality of life.

Endoanal ultrasound (where an ultrasound probe is inserted directly into the back passage) is the gold standard diagnostic tool to detect OASIs. It is however not available in most obstetric units. Transperineal ultrasound (where an ultrasound probe is placed on the perineum)(TPUS) in contrast is available in most obstetric units and therefore we wish to determine whether TPUS in addition to a routine clinical examination will increase the detection rate of OASIs.

Anal incontinence can also occur if the anal sphincter are not repaired adequately. Therefore we want to investigate whether the use of TPUS immediately after primary repair of OASIs is an useful tool to minimise an inadequate repair.

The other aim of the study is to look at changes that occur to the pelvic floor muscles during labour by ultrasound. It is known that certain muscle changes may lead to urinary incontinence and pelvic organ prolapse. However limited studies have evaluated the natural history of the pelvic floor muscles in labour. We therefore wish to perform a transperineal ultrasound each time the midwife or doctor caring for the woman in labour decides the woman in labour needs a vaginal examination. This will provide important information regarding changes that occur to the muscles of the pelvic floor during normal labour.

References:

1)Byrd L,Hobbiss J,Tasker M. Is it possible to predict or prevent third degree tears? Colorectal Dis 2005;7:311-8.

ELIGIBILITY:
Inclusion Criteria:

* women who are undergoing their first vaginal delivery
* 37 weeks of gestation or more
* a singleton pregnancy
* cephalic presentation
* maternal age 18 years old or more and being able to read and understand English.

Exclusion Criteria:

* Exclusion criteria are those who do not fit in the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who delivered vaginally or by caesarean section.
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic test accuracy of three dimensional and transperineal ultrasound (TPUS) for diagnosing Obstetric Anal Sphincter injurieS (OASIS) | immediately Postpartum
  To calculate the diagnostic test characteristics (e.g sensitivity, specificity, positive predictive value, negative predictive value) to enable comparison of 3D TPUS assessment with clinical examination findings of the anal sphincter following vaginal delivery

SECONDARY OUTCOMES:
Prevalence of Levator Ani Muscle Injury in women who delivered vaginally and by caesarean section | during first and second stage of labour, immediately Postpartum, 3 months Postpartum and 10-12 weeks Postpartum (in women who deliver vaginally)
  To calculate the prevalence of levator ani muscle avulsion in women after caesarean section and vaginal delivery.
Levator ani muscle hiatus area (cm2) | during first and second stage of labour, immediately Postpartum, 3 months Postpartum and 10-12 weeks Postpartum (in women who deliver vaginally)
  Levator hiatal dimensions can be determined on three dimensional transperineal ultrasound by identifying the plane of minimal dimensions.
Fetal head position | during first and second stage of labour
  Fetal head position is assessed by clinical examination and transabdominal ultrasound. The possible outcomes of both assessments are occiput anterior, occiput posterior or occiput transverse.
Fetal head station assessed by clinical examination | during first and second stage of labour
  Fetal head station is assessed by clinical examination. The fetal station is the relationship of the presenting part to the ischial spines. It is measured in centimetres above or below the ischial spines (+2,+1,0,-1 or -2).
Fetal head station assessed by transperineal ultrasound | during first and second stage of labour
  Transperineal ultrasound is used to assess fetal head station by measuring the angle of progression. Angle of progression is the angle between the longitudinal axis of the pubic bone and a line joining the lowest edge of the pubis to the fetal skull contour.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Woon Wong, MBBS, Principal Investigator — University Hospital Lewisham
Locations (1):
- University Hospital Lewisham, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03912142/Prot_000.pdf